CLINICAL TRIAL: NCT05904158
Title: Effects of Platelet-Rich Fibrin on Knee Muscle Strength and Function in Patients With Anterior Cruciate Ligament Reconstruction
Brief Title: Effects of Platelet-Rich Fibrin in Patients With Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, SERDAR DEMIRCI, Dr. Fzt. Serdar Demirci (Director of the study), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-18-2060
Record Dates: First submitted 2023-05-27; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Effects of Platelet-Rich Fibrin on Knee Stability and Knee Function
Keywords: Anterior cruciate ligament; platelet-rich fibrin; return to play

STUDY DESIGN:
Intervention Model Description: Randomised controlled design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Group (Experimental): Patients in this group, received PRF application during the standard ACL reconstruction surgery
  Interventions: Biological: Platelet-Rich Fibrin during Standard ACL reconstruction surgery
- Control Group (Active Comparator): Patients in this group received a standard ACL reconstruction surgery without any other intervention.
  Interventions: Other: Standard ACL reconstruction surgery

INTERVENTIONS:
Biological: Platelet-Rich Fibrin during Standard ACL reconstruction surgery — Plateleth-rich fibrin was obtained from patients own blood (40 cc) and applied to the tunnels which were drilled for ACL graft
  Arms: PRF Group
Other: Standard ACL reconstruction surgery — This was a control group where patients received Standard ACL reconstruction surgery
  Arms: Control Group

SUMMARY:
The study was conducted to investigate the effects of platelet-rich fibrin on knee stability, knee muscle strength and knee function in patients with ACL reconstruction. Thirty patients with ACL reconstruction were included to the study and randomly divided into two groups. Patients were assessed preoperative and at the postoperative 1-year.

DETAILED DESCRIPTION:
The study was conducted yo investigate the effects of platelet-rich fibrin (PRF) on the knee stability and function in patients with anterior cruciate ligament (ACL) reconstruction. Thirty patients with ACL reconstruction were included to the study and randomly divided into two groups (PRF group and control group). Hamstring tendon autograft was used in all patients for the reconstruction of the teared ACL. A standardized postoperative rehabilitation program was applied to all patients. Patients' knee stability, knee muscle strength and knee function were assessed preoperatively and one-year postoperatively. Knee stability was assessed using KT-2000 Knee Arthrometer. Quadriceps femoris and hamstring muscle strength measurements were conducted with an isokinetic dynamometer at 60˚/sec and 180˚/sec angular velocities. One Leg Hop (OLH) and Y-Balance tests, and International Knee Documentation Committee (IKDC) were used to evaluate the knee function.

ELIGIBILITY:
Inclusion Criteria:

* Being isolated ACL reconstruction,
* Being between the ages of 18-45 years,
* Performing sports recreationally or professionally

Exclusion Criteria:

* Having previous knee surgery,
* Having systematic disease,
* Having multiple ligament injury on the knee or additional cartilage injuries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Changes in the Knee Laxity | Preoperatively ans one year postoperatively
  Knee laxity was measured using Kneelax-3 Knee arthrometer

SECONDARY OUTCOMES:
Changes in the Knee Muscle Strenght | Preoperatively ans one year postoperatively
  Qudriceps and hamstring muscle strength were measured using an isokinetic dynamometer
Changes in the Knee Function | Preoperatively and one year postoperatively
  Knee function was assessed with one leg hop (OLH) test and Y-Balance tests

IPD SHARING:
Plan to Share IPD: No